CLINICAL TRIAL: NCT07055737
Title: Effectiveness of Aerobic and Barre Exercises on Psychological Well-being Among Postpartum Females
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall20/1017
Record Dates: First submitted 2025-06-28; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Psychology, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supervised aerobic activities (Experimental)
  Interventions: Combination Product: supervised aerobic activities
- Barre group performed light warm-up (Experimental)
  Interventions: Combination Product: Barre group performed light warm-up

INTERVENTIONS:
Combination Product: supervised aerobic activities — Participants performed supervised aerobic activities including warm-up (15 min), brisk walking, jogging, or cycling (30 min), squats on exercise ball (10 min), and cool down (5 min). Sessions were conducted three times a week
  Arms: supervised aerobic activities
Combination Product: Barre group performed light warm-up — Barre group performed light warm-up (15 min), lower abdominal crunches, leg raises, wall push-ups, and planks (3 sets each), followed by cool-down stretches (5 min). Sessions were conducted three times a week.
  Arms: Barre group performed light warm-up

SUMMARY:
This study is a single-blinded randomized controlled trial designed to compare the effectiveness of aerobic exercises and Barre exercises in improving psychological well-being among postpartum females. A total of 44 participants aged between 18-35 years, within 6-12 weeks postpartum, were randomly assigned to two groups: Group A received aerobic exercises while Group B received Barre training.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18-35 years
* Postpartum duration of 6-12 weeks
* Experiencing symptoms of depression, anxiety, or mood disturbance

Exclusion Criteria:

* History of neonatal death
* More than 3 miscarriages
* Diagnosed psychiatric conditions
* Pre-eclampsia, gestational diabetes, or cardiovascular illness
* Currently on psychiatric medications

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scal | 6 Month
  EPDS (Edinburgh Postnatal Depression Scale): 10 items; scored 0-30; higher scores indicate greater depression risk. Score >12 considered clinically significant.
Generalized Anxiety Disorder Scale | 6 Months
  GAD-7 (Generalized Anxiety Disorder Scale): 7 items; scored 0-21; higher scores indicate greater anxiety. Score ≥10 suggests moderate/severe anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No